CLINICAL TRIAL: NCT04009694
Title: Does a High BMI Affect Supervised Pelvic Floor Muscle Training for Improving Symptoms in Women With Various Stages of Pelvic Organ Prolapse?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Salford (Other)
Responsible Party: Principal Investigator, Rebecca Whittle, Rebecca Whittle BSc Hons. Specialist Pelvic Health Physiotherapist, University of Salford
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: USalford1
Record Dates: First submitted 2019-07-02; First posted 2019-07-05 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Pelvic Organ Prolapse; Uterine Prolapse; Anterior Wall; Prolapse, Vaginal; Posterior Wall; Prolapse, Vaginal; Cystocele; Rectocele; Vault Prolapse, Vaginal
Keywords: Pelvic floor muscle training; pelvic physiotherapy; pelvic floor exercises
MeSH Terms: conditions — Pelvic Organ Prolapse; Uterine Prolapse; Prolapse; Cystocele; Rectocele

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pelvic Floor Muscle Training (Experimental): Sixteen weeks of supervised pelvic floor muscle training with a specialist physiotherapist.
  Participants will be assessed at weeks 0 / 4 / 10 & 16 and the outcome measures will be recorded at week 0 & week 16.
  During each assessment, participants will be educated regarding the anatomy of pelvic organ prolapses and the pelvic floor muscles. They will be taught how to contract their pelvic floor, offered a vaginal examination, given a personalised pelvic floor muscle training programme (including the Knack) - up to a ten second hold long contractions (x 10 repitations) and up to 10 quick contractions. They will also be taught a sub max contraction for up to 30 seconds, offered lifestyle management advice including avoiding heavy lifting or straining. A leaflet explaining the aforementioned information will also be provided at the initial assessment.
  Interventions: Other: Pelvic Floor Muscle training

INTERVENTIONS:
Other: Pelvic Floor Muscle training — Sixteen weeks of supervised pelvic floor muscle training with a specialist physiotherapist

SUMMARY:
The trial design is a quasi-experimental cohort trial that includes women referred for pelvic organ prolapse specific physiotherapy.

Candidates will be selected via a convenience sampling method from four physiotherapy outpatient departments at a NHS trust within Greater Manchester. The data collection occurred in January-June 2019 and ethical approval was granted by School Research Ethics, University of Salford.

Treatment aims to ensure there is respect for their autonomy, treatment is fair (Justice), no harm is done to the participant (nonmaleficence) and treatment benefits the participants (beneficence).

Participants are required to complete a consent form prior to their initial session. To ensure methodological quality, the STROBE guidelines will be followed to make certain all apt information required is reported to allow for replication of the intervention.

The trial aims to include (n=60) women with a diagnosed pelvic organ prolapse. They are required to complete 16 weeks of supervised pelvic floor exercises with a specialist physiotherapist as documented within the most recent NICE guidelines.

The outcome measures used will be the Pelvic Organ Prolapse symptom score (POPSS) and this will be documented before and after the 16 week period.

Along side the POPSS, the patients body mass index and severity of pelvic organ prolapse will also be recorded and the results of this will be correlated post trial using the relevant data analysis testing methods.

ELIGIBILITY:
Inclusion Criteria:

* Gynaecologist diagnosed women with a mild / moderate or severe pelvic organ prolapse
* >18 years old

Exclusion Criteria:

* Unwilling or unable to provide informed consent (opt out of treatment)
* Unable to contract the pelvic floor muscles (determined by the treating physiotherapist)
* History of Pelvic cancer / or radiotherapy treatment within three months,
* Neurological or psychiatric disorders,
* Untreated urinary tract infections,
* Pregnant or planning to become pregnant or given birth within the past year,
* Recent vaginal surgery within twelve weeks or evidence of genital oedema,
* Suspected infection or fragility of the genital area As indicated by the referral source or patient reported at the initial assessment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pelvic organ prolapse is a condition exclusive to women
Enrollment: 60 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-09-01 (Estimated); Study Completion 2019-09-10 (Estimated)

PRIMARY OUTCOMES:
Pelvic Organ Prolapse Symptom Score (POPSS) | sixteen weeks
  The POPSS is a patient-reported Outcome Measure consisting of seven POP symptom specific items, each with a five-point Likert response set (0 = never, 1 = occasionally, 2 = sometimes, 3 = most of the time and 4 = all of the time). The minimum score is 0 which would indicate that the pelvic organ prolapse in a-symptomatic and the maximum score for the POPSS is 28 which would indicate higher severity in pelvic organ prolapse symptoms. In addition, the women select a specific symptom which is most bothersome for them.

CONTACTS AND LOCATIONS:
Overall Officials: Nicky Spence, PhD, Study Chair — University of Salford
Locations (1):
- National Health Service, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes